CLINICAL TRIAL: NCT01298713
Title: Phase 2 Study Assessing the Tolerance and Efficacy of Tamoxifen Alone Versus the Association Tamoxifen-RAD001 (Everolimus) in Patients With Anti-aromatase Resistant Breast Metastatic Cancer
Brief Title: Tamoxifen-RAD001 Versus Tamoxifen Alone in Patients With Anti-aromatase Resistant Breast Metastatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAMRAD; EUDRACT 2006-004332-79
Record Dates: First submitted 2011-02-16; First posted 2011-02-18 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Breast Neoplasms; mTor Protein
Keywords: Hormonoresistance; tamoxifen; Previously received anti-aromatase treatment; mTor inhibitor
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Tamoxifen 20mg/d
  Interventions: Drug: Tamoxifen
- B (Experimental): Tamoxifen 20mg/d + RAD001 10mg/d
  Interventions: Drug: Tamoxifen; Drug: Everolimus

INTERVENTIONS:
Drug: Tamoxifen — 20mg daily (1 cap) until unbearable toxicity or progression
Drug: Everolimus — 10mg daily (2 caps of 5mg) until unbearable toxicity or progression
  Other Names: RAD001
  Arms: B

SUMMARY:
Tamoxifen is a classical treatment for breast metastatic cancer after 3rd generation anti-aromatase hormonotherapy in adjuvant or in metastatic line. The Tamoxifen efficacy is lowered by the hormonoresistance mechanisms due to the primary use of the anti-aromatases. The Pi3K-AKT-mTor pathway is frequently associated to the hormonoresistance mechanisms. This study is aimed to check if the inhibition of this signal transduction pathway by a synthetic mTor inhibitor (Everolimus) could improve the efficacy of the Tamoxifen.

ELIGIBILITY:
Inclusion Criteria:

* Menopausal female patient aged > 18 years
* Histologically proven breast adenocarcinoma
* ER and/or PR positive receptors and HER2 negative
* previously received first or second line of hormonotherapy for metastatic disease
* previously treated with anti-aromatase in adjuvant and/or in metastatic line
* presence of one or several mesurable or evaluable metastatic lesion(s)
* presence of at least one target lesion not previously irradiated
* ECOG Performance status < 2
* adequate biological values
* patient who has clearly given her consent by signing on informed consent form prior to participation

Exclusion Criteria:

* patient with only local metastatic disease that can be treted by surgery
* uncotrolled brain metastases, pulmonary carcinomatosal lymphangitis, hepatic metastases
* Previous treatment by Tamoxifen unless in adjuvant and terminated more than a year before metastatic relapse
* Patient with a tumor surexpressing HER2 that should be treated by trastuzumab
* Patient that need an immediate local antalgic radiotherapy
* Thrombo-embolism disease
* serious concomitant pathology or uncontrolled that is susceptible to compromise the participation in the study
* history of another malignancy within past 5 years that could confound diagnosis or staging of breast cancer (with the exception of in situ cacinoma of the cervix or adequately treated basel cell carcinoma of the skin) and cancers cured for at least for 5 years
* patient with an history of significant cardiovascular impairment (congestive heart failure> NYHA grade II, unstable angina or myocardial infraction within the past six months or serious cardiac arrhythmia)
* patient with any medical or psychiatric condition that, in the opinion of the Principal Investigator, would preclude her from participating in this study
* patient with a known allergy to one or several of the study compounds
* patients who may not be regularly available due to geographical, social or family reasons
* history of renal, hepatic or metabolic pathology that could preclude with metabolism or elimination of the study product
* deficiencies of the upper intestinal tract, malabsorption syndrome
* patient who is pregnant, breast-feeding or using inadequate contraception
* Treatment with experimental drugs (mTor inhibitor or tyrosin kinase inhibitor)
* Patient treated with molecules that interfer with isoenzyme CYP3A

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2018-09-12 (Actual)

PRIMARY OUTCOMES:
Clinical benefit at 24 weeks | 42 months

SECONDARY OUTCOMES:
Partial and complete response per RECIST | 42 months
Qualitative and quantitative toxicities | 24 months
Overall survival | 42 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Hotel Dieu, Paris, France

REFERENCES:
- [Derived] Treilleux I, Arnedos M, Cropet C, Wang Q, Ferrero JM, Abadie-Lacourtoisie S, Levy C, Legouffe E, Lortholary A, Pujade-Lauraine E, Bourcier AV, Eymard JC, Spaeth D, Bachelot T. Translational studies within the TAMRAD randomized GINECO trial: evidence for mTORC1 activation marker as a predictive factor for everolimus efficacy in advanced breast cancer. Ann Oncol. 2015 Jan;26(1):120-125. doi: 10.1093/annonc/mdu497. Epub 2014 Oct 31. PMID 25361980